CLINICAL TRIAL: NCT00373997
Title: Role of Esophageal and Laryngeal Biopsies in Suspected Laryngopharyngeal Reflux
Brief Title: Esophageal and Laryngeal Tissue Changes in Patients Suspected of Having Laryngopharyngeal Reflux
Acronym: biopsy I
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Michael Vaezi, Principal Investigator, Vanderbilt University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 060725
Record Dates: First submitted 2006-09-05; First posted 2006-09-08 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2011-03

CONDITIONS: Larynx Disease; Gastroesophageal Reflux
MeSH Terms: conditions — Laryngeal Diseases; Gastroesophageal Reflux | interventions — Endoscopy, Digestive System; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Esophageal and Laryngeal biopsies — one day procedure
  Other Names: esophagogastroduodenoscopy
Procedure: egd with biopsy — standard of care procedure with biopsy
  Other Names: esophagogastroduodenoscopy

SUMMARY:
The purpose of the study is to determine whether patients with suspected Laryngopharyngeal reflux have inflammation and ultrastructural injury on their laryngeal biopsies.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) has been implicated, in part, as the cause of various laryngeal signs and symptoms (1-7). This is often termed reflux laryngitis, ear, nose, and throat (ENT) reflux, or laryngopharyngeal reflux (LPR). GERD was first described to be a causative agent in developing contact ulcers of the larynx (8), and since this early report other routinely observed laryngeal signs are now attributed to LPR. These include laryngeal edema/erythema, vocal cord granulomas and polyps, posterior cricoid cobblestoning, interarytenoid changes, and subglottic stenosis. In addition, patient symptoms attributed to LPR include hoarseness, sore or burning throat, chronic cough, throat clearing, globus, nocturnal laryngospasm, otalgia, post-nasal drip, and dysphagia.

GERD occurs in 7% - 25% of the population on a daily or monthly basis, respectively (9). It is estimated that up to 10% of patients presenting to ENT physicians do so because of complaints that are thought to be related to LPR (2).

The current management of patients with suspected LPR complaints include either 1. empiric therapy using proton pump inhibitors (PPI's) or 2. Ambulatory 24hour pH monitoring to test for GERD before beginning treatment. Because of the uncertainty and subjectivity of the ENT laryngeal examination in diagnosing LPR, both algorithms fall short of ideal in treating these patients. In a recent review of the literature, remarkably, up to 50% of patients with laryngoscopic signs suggesting LPR do not respond to aggressive acid suppression and do not have abnormal esophageal acid reflux values on pH testing (10). Yet, in this subset of patients LPR continues to be implicated as the probable etiology of the patients laryngeal signs and symptoms.

Calabrese, et al. recently looked at the reversibility of GERD related ultrastructural alterations in the esophagus using a PPI. Lower esophageal biopsies were analyzed with electron microscopy (EM) for ultrastructural alterations attributed to GERD; that is, dilation of intracellular spaces. Patients were then treated with a PPI and re-biopsied for analysis of any changes of healing that may have occurred in these ultrastructural alterations. Not surprisingly, the ultrastructural alterations showed complete recovery (reduction of dilated intracellular spaces) after treatment with a PPI. Additionally resolution of patients symptoms coincided with recovery of ultrastructural alterations (11). No such biopsies looking for LPR related changes in the larynx have ever been performed in human subjects.

In sum, LPR is an extremely subjective diagnosis, in which nearly half of all patients do not have an abnormal 24hr pH study, nor do they respond to the standard GERD therapy of acid suppression. Finding an alternative objective criterion for GERD induced laryngitis would be an important clinical discovery. To date, there are no data on microscopic changes in the larynx of patients suspected of having LPR.

In sum, LPR is an extremely subjective diagnosis, in which nearly half of all patients do not have an abnormal 24hr pH study, nor do they respond to the standard GERD therapy of acid suppression. To date, there is no microscopic evidence of laryngeal damage caused by LPR.

ELIGIBILITY:
Inclusion Criteria

* GERD 1. Documented erosive esophagitis (Patients will be newly diagnosed with esophageal erosion at initial visit via esophagogastroduodenoscopy [EGD]) 2.Patients with non-erosive esophagitis who have been responsive to PPI
* LPR 1. Diagnosed via Head & Neck Institute endoscopists (i.e. patients will be newly diagnosed at initial visit via laryngoscopy)
* Controls

  1. No complaints or history of heartburn, acid regurgitation, atypical chest pain
  2. Never been seen by GI or ENT for related symptoms
  3. No prior therapy for GERD
  4. Have a medical condition other than reflux for which they need to undergo EGD. These conditions can be diarrhea, peptic ulcer disease, malabsorption, anemia, and dysphagia.

Exclusion Criteria

* Age < 18yrs
* Pregnancy
* Patients with contra-indications for EGD
* Use of antacid (PPI, H2RB) within last 30 days
* Use of any/all medications affecting gastrointestinal motility
* Known history of: Barrett's esophagus, Peptic stricture, Pyloric stenosis, Gastric resection
* Patients unable to give informed consent
* Patients unable to comply with follow-up
* Contraindications to biopsy: Taking anticoagulants other than aspirin (Coumadin, Plavix) or allergies to local anesthetic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2006-09; Primary Completion 2009-03 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Dilation of intracellular spaces at the beginning of the study | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Vaezi, MD, PhD, MS epi, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Endoscopy Lab, TVC 1410, Nashville, Tennessee, United States